CLINICAL TRIAL: NCT02663609
Title: Retrospective Chart Review Study of Korlym for the Treatment of ACTH Independent Cushing's Syndrome
Acronym: RE-KLAIM
Status: Completed | Type: Observational
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: C1073-450
Record Dates: First submitted 2016-01-08; First posted 2016-01-26 (Estimated); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Cushing's Syndrome
Keywords: Cushing's Syndrome; Mifepristone; Adrenal; Retrospective; Chart Review
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: No intervention — No treatment (intervention) was administered.

SUMMARY:
Chart review study to collect patient data from medical charts of patients who have been treated with Korlym® for the treatment of ACTH independent adrenal Cushing's Syndrome.

DETAILED DESCRIPTION:
A retrospective, multi-center, chart review study to collect patient data from medical charts of patients who have been treated with Korlym® for the treatment of ACTH independent adrenal Cushing's Syndrome. Treatment with Korlym® will be a minimum 3 months in duration with follow-up of a minimum 3 months. Only sites that have been identified to have patients appropriate for this protocol will be invited to participate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ACTH independent endogenous Cushing's Syndrome
* Available adrenal imaging prior to being treated with Korlym®
* Treated with Korlym® and followed for at least 3 months (follow-up data should be available)

Exclusion Criteria:

* Diagnosed with adrenocortical carcinoma
* Participant in any clinical trial(s) during the observational period

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ACTH Independent Cushing's Syndrome patients treated with Korlym® mifepristone) as standard of care in clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

PRIMARY OUTCOMES:
Drug Utilization Patterns as assessed by chart review | up to 4 years
  The retrospective review would analyze the drug utilization patterns of patients treated with Korlym

SECONDARY OUTCOMES:
Clinical Outcomes as assessed by chart review | up to 4 years
  The retrospective review would analyze outcomes measures (vitals, clinical assessments, etc) in patients treated with Korlym

IPD SHARING:
Plan to Share IPD: No